CLINICAL TRIAL: NCT06973109
Title: Investigating the Efficacy of Romosozumab in Augmenting Bone Density and Muscle Mass to Enhance the Outcomes of Spine Surgery
Brief Title: Romosozumab Effects on Bone Density, Muscle Mass, and Spine Surgery Outcomes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nitin Agarwal (Other)
Collaborators: Amgen (Industry); Beckwith Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Nitin Agarwal, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY24090048; BECKW 12879 (Other Grant/Funding Number: Beckwith Institute); 2024YIRGA (Other Grant/Funding Number: AO Spine)
Record Dates: First submitted 2025-05-02; First posted 2025-05-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Osteoporosis, Post-menopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — romosozumab; Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Romosozumab + Placebo Alendronate (Experimental): Participants will receive monthly subcutaneous injections of romosozumab (210 mg, one injection per arm) for 12 months, along with weekly oral placebo alendronate. Surgery will be performed 3 months after treatment initiation. DXA and CT scans will assess bone density and muscle mass. Functional outcomes will be evaluated via PROMs at baseline and follow-up.
  Interventions: Drug: Romosozumab; Drug: Placebo Alendronate
- Alendronate + Placebo Romosozumab (Active Comparator): Participants will receive weekly oral doses of alendronate (70 mg) and monthly subcutaneous placebo injections mimicking romosozumab. Surgery will occur after 3 months of treatment. Bone density, muscle mass, and functional outcomes will be assessed similarly to the experimental arm.
  Interventions: Drug: Alendronate (Fosamax); Drug: Placebo Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Monthly subcutaneous injection (210 mg total dose) administered as two separate 105 mg injections, one per arm. Administered for 12 months to female patients ≥65 years undergoing spine surgery.
  Other Names: Evenity
  Arms: Romosozumab + Placebo Alendronate
Drug: Alendronate (Fosamax) — Weekly oral dose (70 mg) administered for 12 months. Used as active comparator in control arm of study.
  Other Names: Fosamax
  Arms: Alendronate + Placebo Romosozumab
Drug: Placebo Romosozumab — Monthly subcutaneous injections mimicking romosozumab in appearance and administration schedule. Administered to control group.
  Arms: Alendronate + Placebo Romosozumab
Drug: Placebo Alendronate — Weekly oral placebo pill mimicking alendronate. Administered to treatment group.
  Arms: Romosozumab + Placebo Alendronate

SUMMARY:
The goal of this clinical trial is to learn if romosozumab (Evenity) can improve bone and muscle health in postmenopausal women with osteoporosis who are undergoing lumbar spine surgery. The main questions it aims to answer are:

* Does romosozumab improve bone strength and reduce the risk of complications during and after spine surgery?
* Does romosozumab increase muscle mass and help patients recover better from surgery?

Researchers will compare romosozumab (a monthly injection) to alendronate (a weekly pill), both approved treatments for osteoporosis, to see which is more effective in this surgical setting. Participants will:

* Be randomly assigned to receive romosozumab or alendronate
* Take standard vitamin supplements and receive a one-time dose of zoledronic acid near the end of the study
* Attend five study visits over about 12 months
* Undergo bone scans, muscle imaging, and complete health questionnaires before and after surgery

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal female
* Diagnosed with osteoporosis (T-score ≤ -2.5).
* Scheduled for or planning posterior lumbar fusion for degenerative disease, at least 3 months in the future.
* Able to provide informed consent.

Exclusion Criteria:

* History of prior spinal surgery.
* Male sex.
* Current or prior use of osteoporosis medications within the past 3 years.
* Current use of anabolic agents other than romosozumab.
* Current use of androgen receptor (AR) modulators, such as testosterone replacement therapy or selective androgen receptor modulators (SARMs).
* Severe renal impairment (eGFR < 30 mL/min/1.73m²).
* Known hypersensitivity to romosozumab, alendronate or zoledronic acid.
* Severe spinal deformity.
* Active malignancy or history of malignancy within the past 5 years.
* Any secondary cause of decreased BMD (e.g., hyperparathyroidism).
* Stroke or myocardial infarction in the past year.
* Planned fusion involving more than 4 levels.
* Uncorrected hypocalcemia and/or hypovitaminosis D
* Esophageal abnormalities

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-17 (Estimated); Primary Completion 2027-01-26 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Hounsfield Units (HU) at L1 Vertebra | Baseline, 3 months post-op, and 9 months post-op
  This measure assesses changes in vertebral bone quality by measuring Hounsfield Units (HU) at the L1 vertebra via CT scans. HU values will be compared from baseline to post-treatment between the romosozumab and alendronate groups to evaluate bone density improvement.
Change in Vertebral Bone Mineral Density (BMD) at L1 | Baseline, 3 months post-op, and 9 months post-op
  This measure evaluates the efficacy of romosozumab in improving vertebral bone density in older adults undergoing spine surgery. BMD will be measured using DXA scans of the total hip and compared from baseline to post-treatment between the romosozumab and alendronate groups.

SECONDARY OUTCOMES:
Change in L3 skeletal muscle index (L3 SMI) | Baseline, 3 months post-op, and 9 months post-op
  This measure assesses the impact of romosozumab on muscle mass in patients undergoing spine surgery. L3SMI will be calculated from axial CT scans at the L3 vertebral level, normalized by patient height squared. Changes from baseline will be compared between treatment and control groups.
Change in Oswestry Disability Index (ODI) | Baseline and 9 months post-op
  This measure evaluates change in patient-reported disability related to lower back pain using the ODI. Scores range from 0 to 100, with higher scores indicating greater disability.
Change in Visual Analog Scale (VAS) for Pain | Baseline and 9 months post-op
  This measure evaluates change in pain intensity using the VAS, which ranges from 0 (no pain) to 10 (worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Agarwal, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center (UPMC) - Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) collected during the trial that underlies published results will be shared, including de-identified data on demographic variables, dual-energy X-ray absorptiometry (DXA) bone mineral density (BMD) measurements, Hounsfield unit (HU) values from CT scans, L3 skeletal muscle index, radiographic fusion outcomes, hardware complication data, and patient-reported outcomes (ODI and VAS scores). Data will be made available to other qualified researchers upon reasonable request following publication of primary results, contingent on IRB approval and data use agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information will be available beginning 12 months after publication of the primary results and will remain available for 5 years thereafter.
Access Criteria: Qualified researchers with a methodologically sound proposal may request access to the data by contacting the study principal investigator. Requestors will need to complete a data use agreement. Data will be provided via a secure online platform after IRB approval and review of the request by the study team.
URL: https://www.scoli.org/